CLINICAL TRIAL: NCT02992041
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Dose Finding Study to Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injections for Post-Operative Pain Following Laparoscopic Colorectal Surgery
Brief Title: Evaluate the Analgesic Efficacy and Safety of VVZ-149 Injections for Post-Operative Pain Following Laparoscopic Colorectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVZ149-POP-P2-US002
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower dose VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Higher dose VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 Injections — IV infusion of 900 or 1100 mg of VVZ-149
  Other Names: Opiranserin Injections
  Arms: Higher dose VVZ-149 Injections; Lower dose VVZ-149 Injections
Drug: Placebo — IV infusion of 0 mg of VVZ-149
  Arms: Placebo

SUMMARY:
The purpose of this phase 2 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections. The study is designed as randomized, double-blind, parallel, placebo-controlled study.

DETAILED DESCRIPTION:
VVZ-149 is a dual antagonist of GlyT2 and 5HT2A. GlyT2 blockage increases inhibitory synaptic transmission by glycine in the spinal cord, resulting in a reduction of pain transmissions to the brain. 5HT2A blockage decreases descending serotonergic facilitatory modulation on pain transmission by the brain and reduces nociceptor activation in peripheral nerves, which are primary sources of pain in post-surgical pain. VVZ-149 has been shown to have comparable efficacy to morphine in well controlled (blind, complete randomization with a positive control) animal studies using rat models of post-operative pain and formalin-induced pain. The PK/PD study in animals indicates that therapeutic plasma concentration in human subjects will be 600-1,900 ng/ml. A clinical Phase 1 study performed in healthy subjects has shown no clinically significant adverse events up to a plasma concentration level of 3,261 ng/ml other than brief symptoms of mild nausea or dizziness, and mild somnolence when the plasma exposure level is more than 2,000 ng/ml. A clinical Phase 2 study performed in laparoscopic gastrectomy patients showed that patients who received VVZ-149 had reduced opioid consumption after surgery compared to those who received placebo, without any significant drug-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing planned laparoscopic colorectal surgery.
* Ability to provide written informed consent.
* Ability to understand study procedures and communicate clearly with the investigator and staff.
* American Society of Anesthesiologists (ASA) risk class of I to III.

Exclusion Criteria:

<Surgical Factors>

* Emergency or unplanned surgery.
* Repeat operation (e.g., previous surgery within 30 days for same condition).
* Cancer-related condition causing preoperative pain in site of surgery.
* Surgical duration (from incision to end of closure) > 5 hours.

<Subject Characteristics>

* Women with childbearing potential (age 18-55) must undergo blood pregnancy test at screening and then a urine pregnancy test preoperatively on day of surgery. Women with a positive pregnancy test will be excluded. Women of childbearing potential must agree to use at least one effective contraceptive method upon enrollment and for 30 days following the last dose of the investigational product.
* Women who are pregnant or breastfeeding.
* Chronic pain diagnosis (e.g., ongoing pain at baseline with NRS ≥ 4/10).
* Unstable or poorly controlled psychiatric condition (e.g., untreated PTSD, anxiety, or depression) Subjects who take stable doses of antidepressants and anti-anxiety drugs, or procedure-related anti-anxiety drugs may be included.
* Unstable or acute medical condition (e.g., unstable angina, congestive heart failure, renal failure, hepatic failure, AIDS).
* Body weight under 55 kg.

<Drug, Alcohol, and Pharmacological Considerations>

* Renal or hepatic impairment.
* History of alcohol, opiate or other drug abuse or dependence within 12 months prior to Screening (TICS alcohol/drug screen will be performed at Screening).
* Ongoing or recent (within 30 days prior to surgery) use of opioids or antipsychotics. However, subjects who receive procedure-related opioids (i.e., for a preoperative colonoscopy) may be included.
* Alcohol consumption within 24 hours of surgery.
* Use of nonsteroidal anti-inflammatory drugs (NSAIDs) or acetaminophen within 24 hours of surgery. Exception: use of aspirin for cardiovascular prophylaxis is acceptable.
* Use of herbal agents or nutraceuticals (i.e., chaparral, comfrey, germander, jin bu huan, kava, pennyroyal, skullcap, St. John's wort, or valerian) within 7 days prior to surgery.

<Anesthetic and Other Exclusion Considerations>

* Use of neuraxial or regional anesthesia related to the surgery.
* Use of local anesthetic wound infiltration > 20 ml of 1% lidocaine
* Use of ketamine, gabapentin, pregabalin, or lidocaine (>1 mg/kg) intra or peri-operatively, or within 24 hours of surgery.
* Subjects with known allergies to hydromorphone.
* Subjects who received another investigational drug within 30 days of scheduled surgery.
* Subjects who have long PR (>200 msec) or prolonged QTc (> 450 msec for males and > 470 msec for females) at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC) of Pain Intensity | 0hr=start of PCA, 1hr and 2 hours
  area under the curve (AUC) of Pain Intensity using Numeric Pain Rating Scale (NRS, 0-10 at rest) measured up to 2 hours post-initiation of PCA

SECONDARY OUTCOMES:
Opioid Consumption up to 24 hours post-dosing of study drug | 0-2, 2-4, 4-6, 6-8, 8-10, 10-12, and 12-24 hours
  Total amount of hydromorphone (including rescue doses) consumption up to 24 hours after starting PCA
Pain Intensity (Numeric Pain Rating Scale, NRS) | 0, 1, 2, 4, 6, 8, 10, 12, and 24 hours
  Pain Intensity (NRS at rest) measured up to 24 hours post-initiation of PCA
Global measurement of subject satisfaction with study medication | 8 and 24 hours post-initiation of PCA
  Global assessment of subject satisfaction with analgesic management using a 5-point scale (0-4)
Richmond Agitation Sedation Scale (RASS) | 0, 1, 2, 4, 6, 8, 10, 12, and 24 hours post-initiation of PCA
Respiratory Depression Assessment | 0, 1, 2, 4, 6, 8, 10, 12, 24 hours post-initiation of PCA and within 10 minutes prior to administering any rescue doses of hydromorphone
Post-Operative Nausea and Vomiting scale (PONV) | 0, 4, 8, 12, and 24 hours post-initiation of PCA

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts